CLINICAL TRIAL: NCT03595241
Title: Prospective, Randomised, Crossover, Controlled, Feasibility Study to Assess the Efficacy of BurstDR Spinal Cord Stimulation (SCS) as a Treatment for Persistent AbdomiNal RefrActory VisCEral PAin Secondary to Chronic Pancreatitis: PANACEA Trial
Brief Title: PANACEA Feasibility Study to Assess the Efficacy of BurstDR Spinal Cord Stimulation (SCS)
Acronym: PANACEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PM15/126
Record Dates: First submitted 2018-06-13; First posted 2018-07-23 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - active treatment (Experimental)
  Interventions: Device: Spinal cord stimulation by implanted device.
- Group B - conservative management (No Intervention)

INTERVENTIONS:
Device: Spinal cord stimulation by implanted device. — Spinal cord stimulation (SCS) protocol from the implanted device. This involves activation of the device for the (SCS) protocol including Burst DR therapy.
  Arms: Group A - active treatment

SUMMARY:
To evaluate the effectiveness of Burst DR stimulation as a treatment for persistent abdominal refractory visceral pain secondary to chronic pancreatitis. Abdominal pain is a main symptom in patients with chronic pancreatitis. Patients have a background constant pain with acute episodes needing admissions. Spinal cord stimulation (SCS) is a recognised treatment for neuropathic pain. This involves placing an electric wire in the spine and the use of electricity to manage the pain. This is a pacemaker for controlling pain. Burst DR stimulation delivers a wave form which mimics the way nerves conduct electrical signals, there are short bursts or spikes of stimulation followed by short periods of rest. The key aims and objectives of this study are to evaluate the efficacy of Burst DR SCS as a treatment for persistent pain secondary to chronic pancreatitis

DETAILED DESCRIPTION:
To evaluate the effectiveness of Burst DR stimulation as a treatment for persistent abdominal refractory visceral pain secondary to chronic pancreatitis. Abdominal pain is a main symptom in patients with chronic pancreatitis. Patients have a background constant pain with acute episodes needing admissions. Spinal cord stimulation (SCS) is a recognised treatment for neuropathic pain. This involves placing an electric wire in the spine and the use of electricity to manage the pain. This is a pacemaker for controlling pain. Burst DR stimulation delivers a wave form which mimics the way nerves conduct electrical signals, there are short bursts or spikes of stimulation followed by short periods of rest. The key aims and objectives of this study are to evaluate the efficacy of Burst DR SCS as a treatment for persistent pain secondary to chronic pancreatitis

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or older (no upper age limit) and willing to provide informed consent
* Participant is able and willing to comply with the follow-up schedule and protocol
* Participants diagnosed with persistent refractory visceral pain secondary to chronic pancreatitis for at least 6 months with or without dermal hyperalgesia or allodynia
* Minimum baseline pain score of 6 on eleven point NRS scale (0-10) for their visceral pain
* Previously tried and failed at least one conservative treatment for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for persistent pain
* Been deemed suitable for the study by the pancreatic or pain MDT
* Total daily dose of opioids equivalent to ≤120mg of Morphine or 50% reduction in opioid dose. If the patients are taking more than this dose, they will be offered a referral to our opioid reduction clinic to achieve the target opioid dose and the baseline opioid will be taken as the dose on referral
* In the investigators opinion, the patient is a suitable candidate for Spinal Cord Stimulation

Exclusion Criteria:

* Female participants of childbearing potential who are pregnant/nursing or plan to become pregnant during the course of the trial
* Escalating or changing pain condition within the past month as evidenced by investigator examination
* Sphlanchnectomy or radiofrequency treatment within the past 6 months
* Currently has an active implantable device including pacemakers, spinal cord stimulator or intrathecal drug delivery system
* In the investigators opinion has an active infection
* Participated in another clinical investigation within 30 days
* Medical co-morbidities that preclude surgical intervention
* Patient is incapable of understanding or operating the patient programmer handset
* Patient is morbidly obese (BMI ≥ 40)
* Participant has a current or previous condition, which will probably require MRI investigation sometime in the following 2 years
* Participant has had a spinal surgical procedure or has spinal pathology that would significantly impede lead implantation at the level planned for implantation
* Participant has another persistent painful condition other than persistent refractory visceral pain secondary to chronic pancreatitis.
* History of alcohol abuse in the last year or IV drug abuse in the last three years.
* No increases of more than 40% from baseline amylase and lipases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of EQ-5D5L Health questionnaire | 1 hour
  Successful completion of EQ-5D5L Health questionnaire leading to a EQ-5D index score (≥0.200) recorded
Numeric Rating Scale (NRS) recording pain severity | 1 hour
  Percentage of change in pain severity recorded on the Numeric Rating Scale (NRS) at four months compared with baseline in both the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain and Interventional Neuromodulation Research Group, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473